# PROJECT TITLE

Effects of a 12-week supervised or home-based multicomponent training program on Psychological, and Physical variables in Fibromyalgia patients.

# LABORATORY/DEPARTMENT

Laboratory of Exercise Science and Sport, Degree Program in Sports Science and Techniques, Department of Translational Biomedicine and Neurosciences (DiBraiN), University of Bari – Aldo Moro

# **EXPERIMENTAL DESIGN**

Interventional

EXPECTED START AND END DATE OF THE PROJECT

March 2025 – June 2025

FUNDS USED FOR THE PROJECT

No

DATE OF THE DOCUMENT

24/04/2025

# INFORMED CONSENT FORM FOR PARTICIPATION IN THE STUDY/RESEARCH PROJECT

Dear Sir/Madam,

You are invited to participate in the research study/project titled "Effects of a 12-week supervised or home-based multicomponent training program on Psychological, and Physical variables in Fibromyalgia patients." In order to make an informed decision, we are providing you with information about the nature of the study, the objectives of the project, and the activities in which you may be involved for the accomplishment of the research goals.

Please read these details carefully before deciding whether to participate in the project. You may ask any questions for clarification and raise any concerns that have not been answered clearly and thoroughly.

If, after reading and understanding all the provided information, you decide to participate in the study, you will be asked to sign and date the attached Informed Consent Form.

Your personal data will be processed as described in the specific privacy notice, in accordance with EU Regulation 2016/679 and Legislative Decree No. 196/2003. This privacy notice and the related request for consent to data processing will be provided to you separately.

**Research title**: Effects of a 12-week supervised or home-based multicomponent training program on Psychological, and Physical variables in Fibromyalgia patients.

CUP Project: N/D Sponsor: N/D

implementing organizations: N/D

# INFORMATION REGARDING PARTICIPATION IN RESEARCH

**OBJECTIVES:** The research project aims to evaluate evaluate the effectiveness of supervised multicomponent training (SMCT) on physiological parameters, physical fitness, mental well-being, and quality of life in subjects with a history of FM, compared to a non-supervised home-based MCT (NSMCT) protocol and a waitlist control group (WLCG). To achieve this objective, the researchers involved in the project aim to collect and analyze data on the estimation of these parameters through physical and psychological tests to be performed before and after the intervention.

#### STUDY/PROJECT ARTICULATION (PHASES AND TIMELINES):

RECRUITMENT PHASE AND COLLECTION OF INFORMED CONSENT (1-3 months)

Presentation to participants: The informed consent will be distributed during the recruitment procedures. The consent will be collected prior to the initial assessments (T0).

RANDOMIZATION PHASE, INITIAL ASSESSMENTS, AND DATA COLLECTION (1-2 weeks)

After recruitment, participants will be randomly assigned to one of the three groups (SMCT, NSMCT, WLCG). Subsequently, initial assessments will be conducted, consisting of motor tests and psychological questionnaires.

#### INTERVENTION PHASE (3 months)

During this phase, participants previously randomly assigned to one of the three groups (SMCT, NSMCT, WLCG), under the supervision of field experts, will begin their activities, specifically:

- SMCT group: Participants will follow a supervised adapted multicomponent training program, which includes aerobic, resistance, and mobility/flexibility exercises;
- NSMCT group: Participants will follow a non-supervised home-based adapted multicomponent training program, which includes aerobic, resistance, and mobility/flexibility exercises;
- WLCG group: Participants will not perform any structured physical activity but will continue with their usual lifestyle. They will be placed on a waiting list, guaranteeing them future participation in adapted physical activity after the intervention period.

# FINAL ASSESSMENT PHASE AND DATA COLLECTION (1-2 weeks)

Within one week after the end of the intervention period, final assessments will be initiated, consisting of motor tests and psychological questionnaires.

**Discussion and Consent Signature:** The research team will clarify any doubts of the participants. Participants will sign the consent form after understanding the details and potential risks. A minimum of 10-30 minutes must be provided per participant.

Estimated Time: 10-30 minutes per participant.

I, the undersigned

**BENEFITS:** Participants will have access to adapted physical activity tailored to their needs, with the aim of improving psychophysical conditions related to mobility, autonomy, and self-efficacy, ultimately enhancing their quality of life, all under the supervision of field experts.

**RISKS:** Participation does not involve any risk or discomfort, except for the rare possibility of traumatic events that may occur during the course of the study.

born in

on

| residing at | stree | et | hereby |
|---|---|---|---|
| | D | ECLARE | |
| that I have read and un | derstood the information | on and wish to particip | eate in the proposed study. |
| | □ I confirm | □ I do not confi | rm |

| <b>SIGNATURE</b> |
|------------------|

A signed copy of the identity document is attached.

For the purpose of informed participation in the research, we invite you to sign the following form, specifying that by signing it, you do not waive any legal rights you are entitled to.

# CONSENT TO PARTICIPATE IN THE RESEARCH

| I declare that: ☐ I have voluntarily decided to participate in the res | search;; |
|---|---|
| $\ \square$ I have received all the information related to the regarding the purpose, procedures, and what is requ | |
| ☐ I have received, read, and understood the do participation in the research," which was provided information for my responsible participation in the research. | d to me, and I have received all the necessary |
| $\hfill \square$<br>I have had the opportunity to ask questions and answers; | have received clear, complete, and satisfactory |
| $\square$ I have been informed about potential risks; | |
| $\square$ I am aware that my participation is voluntary; | |
| $\ \square$ I have been assured that I can withdraw from the negative consequences on the treatment and care I v | • |
| For any doubts or questions, you can contact the <b>Dr</b> Phone 3457687096 | r. Luca Poli |
| Full name of the participant | · |
| Signature of the participant | Date |
| Full name of the person who obtained the consent _ Signature of the research supervisor | Date |
| Full name of any witnesses present | |
| Signature of the witnesses present | <br>Date |

# WITHDRAWAL OF CONSENT

If you wish to withdraw your consent to participate in this research, please indicate with an "X" the desired option among the following:

I withdraw my consent to continue participating in one or more of the following activities (please specify the individual activities for which you wish to exercise the right to withdraw consent):

| • | |
|---|---|
| Full name of the participant Signature of the participant | Date |
| Full name of the person who obtained the consent Signature of the research supervisor | Date |
| Full name of any witnesses present | |
| Signature of the witnesses present | Date |

In case of incapacitated individuals and minors:

# CONSENT DECLARATION FOR THE PROCESSING OF PERSONAL DATA OF THE SUBJECT CONCERNED BY THE PARENT/GUARDIAN/ CURATOR/ SUPPORT ADMINISTRATOR

# PURSUANT TO AND FOR THE PURPOSES OF THE EUROPEAN DATA PROTECTION REGULATION

| I, the un | dersigned | in | | born | on |
|---|---|---|---|---|---|
| | | in | | | |
| in the capacity | | | □ support administrator of | | |
| (name) | in | | _(surname) | , born | |
| | with the provisions of<br>endments and integra | Regulation () | EU) 2016/679 and Legislative Decree having read the "Information on the particle of the partic | 196/2003 ส | |
| | ☐ I co | nsent | ☐ I do not consent | | |
| person concern | ed, including health-r | elated data, f | the research in question - of the person<br>for scientific and statistical research purpose and methods of data | rposes, in | the |
| | ☐ I co | onsent | ☐ I do no consent | | |
| _ | | | articipation in the study in question – or ch activities and to be possibly contact | - | |
| Additionally, | □ I со | nsent | ☐ I do not consent | | |
| other audiovis | | ssary for par | rned (video, audio, and photographic ticipation in the study - for the researce | _ | |
| Date | | | Signature | | |